CLINICAL TRIAL: NCT03930368
Title: Application of Raw Corn Starch on Patients With Unoperated Insulinoma is Helpful to Decrease Risk of Hypoglycemia
Brief Title: Application of Raw Corn Starch on Patients With Insulinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCS-insulinoma
Record Dates: First submitted 2019-04-16; First posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Hyperinsulinemic Hypoglycemia; Insulinoma; Raw Corn Starch
MeSH Terms: conditions — Congenital Hyperinsulinism; Insulinoma

STUDY DESIGN:
Intervention Model Description: In vie of the fact that insulinoma is a rare disease and it will be difficult to enroll enough cases in this study, a prospective single-arm before-and-after study will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervened arm (Experimental): as in a single-arm before-and after study, the only one arm will receive intervention of low GI diet with supplementation of RCS.
  Interventions: Other: low GI diet with regular supplementation of raw corn starch

INTERVENTIONS:
Other: low GI diet with regular supplementation of raw corn starch — Patients will be guided with a low GI diet with 60%~70% of energy from carbohydrates. RCS constituted 30%~50% of daily carbohydrate, and was supplemented as snacks every 4~6 hours (25g per time) especially at night.

SUMMARY:
This will be a prospective single-arm before-and-after clinical trial in which raw corn starch (RCS) will be first applied on patients with unoperated insulinoma. Nutritional intervention with supplementation of RCS will be initiated in 20 patients with suspected insulinoma to improve their hypoglycemia before the surgery. Duration of nutritional intervention, fasting blood glucose, lipid profile, weight change, BMI and other metabolic indices will be recorded and compared before and after the intervention.

DETAILED DESCRIPTION:
Insulinoma is a rare disease which can cause recurrent hyperinsulinemic hypoglycemia, subsequent hyperphagia as well as weight gain. As only 50% ~ 60% of pharmacological therapy (diazoxide, somatostatin, etc) is effective to elevate blood glucose, the nutritional interventions play a role as an important supportive treatment to maintain glycemic stablization and control weight gain before the curative surgery. As the essential management for patients with glycogen storage disease (GSD), the extended release cornstarch has been proved superior to prevent hypoglycemia since 1980s. Its application has elevated GSD patients' quality of life and prolonged their survival. In view of its charicteristic of chronic release in gastrointestinal tract, we will for the first time try to utilize the raw corn starch (RCS) on patients with suspected insulinoma and evaluate its efficacy of improving hypoglycemia in such patients.

This will be a prospective single-arm before-and-after clinical trial. Nutritional intervention with supplementation of RCS will be initiated in 20 patients with suspected insulinoma to improve their hypoglycemia before the surgery. Duration of nutritional intervention, fasting blood glucose, lipid profile, weight change, BMI and other metabolic indices will be recorded and compared before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* having recurrent symptoms of hypoglycemia (blood glucose less than 2.8 mmol/L) which could be relieved by intake of glucose, which condition accords with typical Whipple triad.
* being proved to have abnormally increased secretion of endogeneous insulin at onset of hypoglycemia.
* diagnosis of insulinoma is highly suspected, in view of clinical presentation, laboratory tests and imaging examinations.

Exclusion Criteria:

* severe gastrointestinal dysfunction with intolerance of raw corn starch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
the change of fasting blood glucose | from initiation of nutritional intervention to 2 weeks later, or by the time of curative surgery
  the change of mean fasting blood glucose before and after nutritional intervention
the change of requency of hypoglycemia onset | from initiation of nutritional intervention to 2 weeks later, or by the time of curative surgery
  the change of requency of hypoglycemia onset before and after nutritional intervention
the change of glycated albumin | from initiation of nutritional intervention to 2 weeks later, or by the time of curative surgery
  the change of glycated albumin before and after nutritional intervention

SECONDARY OUTCOMES:
the change of satiety score | from initiation of nutritional intervention to 2 weeks later, or by the time of curative surgery
  the change of self-reported satiety score before and after nutritional intervention. Satiety will be measured using a graphic rating scale that combined verbal descriptors on a scale graded 0-6 (0 = no sensation, 1 = just noticeable/threshold, 2 = very mild, 3 = mild, 4 = moderate, 5 = fullness, 6 = pain)
the change of weight / BMI | from initiation of nutritional intervention to 2 weeks later, or by the time of curative surgery
  the change of weight / BMI before and after nutritional intervention
the change of body fat mass (rate of fat mass) before and after nutritional intervention | from initiation of nutritional intervention to 2 weeks later, or by the time of curative surgery
  the change of body fat mass (rate of fat mass) before and after nutritional intervention, through measurement by bioelectrical impedence analysis
the change of lipid profile (level of total triglycerides, total cholesterol, LDL-C, HDL-C, free fatty acid ) before and after nutritional intervention | from initiation of nutritional intervention to 2 weeks later, or by the time of curative surgery
  the change of total triglycerides, total cholesterol, LDL-C, HDL-C and free fatty acid befor and after nutritional intervention, through measurement by lipid profiles
the change of uric acid | from initiation of nutritional intervention to 2 weeks later, or by the time of curative surgery
  the change of uric acid before and after nutritional intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No